CLINICAL TRIAL: NCT04480892
Title: Fibrinolytic Deficit in Patients With Acute Pulmonary Embolism
Brief Title: Fibrinolytic Deficit in Patients With Acute PE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Loyola University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Amir Darki, Associate Professor, Loyola University
Other Study IDs: 212490
Record Dates: First submitted 2020-06-28; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Acute Pulmonary Embolism; Fibrinolytic Deficit
Keywords: Acute Pulmonary Embolism; Fibrinolytic System; Fibrinolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood samples drawn for clinical evaluation of PE will be collected after analysis complete, de-identified, re-centrifuged, aliquoted, and stored in -80 freezer. Once all 100 patient samples have been collected, samples will be analyzed for fibrinolytic biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fibrinolysis is the body's process that prevents blood clots. The investigators hypothesize that patients presenting with acute pulmonary embolism (PE) or blood clots in the lungs differ in their fibrinolytic deficit phenotype. The investigators aim to use biomarkers directly involved in endogenous fibrinolytic cascade including PAI-1, Alpha-2-Antiplasmin (A2A), TAFI, D-dimer, and Fibrinogen to phenotypically characterize patients presenting with acute PE and to correlate these biomarkers with clinical, echocardiographic, computed tomography (CT), and functional status outcomes.

DETAILED DESCRIPTION:
Patients (n=100) identified by the Pulmonary Embolism Response Team (PERT) suffering from a PE will be identified by the PI. Blood plasma samples from these patients which have been drawn for routine lab tests will be identified and the Sub-I who will pick the samples up from the clinical lab after the routine analysis has been completed. These samples will be de-identified by giving them a study number. These samples will be recentrifuged and aliquoted. Samples will be stored in a -80ᵒC freezer in the Hemostasis & Thrombosis Research Laboratory. When all 100 de-identified samples have been collected they will be analyzed blindly by the technical staff of the hemostasis laboratory for the fibrinolytic parameters PAI-1, Alpha-2-Antiplasmin, TAFI, tPA, D-dimer, Plasminogen, and Fibrinogen. PAI-1 and TAFI will be quantified with an Enzyme Linked-Immuno-Sorbent Assay (ELISA), while A2A is measured using functional assay. PAI-1 is measured as ug/ml, while TAFI and A2A are measured as % of normal controls. Normal controls are derived from pooled normal human plasma from volunteers purchased from outside vendor. Results will be compiled and sent to the PERT team for analysis and correlation withclinical, echocardiographic, computed tomography (CT), and functional status outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 - 90 years
* Patients suffering an acute PE
* Blood collected for clinical evaluation of PE

Exclusion Criteria:

* Blood not collected or not sufficient quantity/quality

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute PE being treated by the PERT.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Plasminogen Activator Inhibitor-1 (PAI-1) | Baseline-Day 1
  Laboratory analysis of blood sample for PAI-1 level
Alpha-2 Antiplasmin level (A2P) | Baseline-Day 1
  Laboratory analysis of blood sample for A2P level
Thrombin Activatable Fibrinolysis Inhibitor (TAFI) | Baseline-Day 1
  Laboratory analysis of blood sample for TAFI level
Tissue plasminogen activator (tPA) | Baseline-Day 1
  Laboratory analysis of blood sample for tPA level
D-dimer | Baseline-Day 1
  Laboratory analysis of blood sample for D-dimer level
Plasminogen | Baseline-Day 1
  Laboratory analysis of blood sample for Plasminogen level
Fibrinogen | Baseline-Day 1
  Laboratory analysis of blood sample for Fibrinogen level
Clinical Presentation Risk Score | Baseline-Day 1
  Based on vital signs (heart rate, blood pressure, oxygen requirements, and labs (CBC, lactate, troponin, and BNP, clinical presentation will be characterized as low, intermediate, or high risk.
Right Ventricular Function | Baseline-Day 1
  Assessed by echocardiography
Pulmonary Artery Pressure | Baseline-Day 1
  Pulmonary Artery Pressure (mmHg) will be measured for patients escalated to endovascular therapies in the cardiac cath laboratory
Cardiac Output | Baseline-Day 1
  Cardiac Output, the volume of blood pumped from the ventricle per heartbeat (mL/min), will be measured for patients escalated to endovascular therapies in the cardiac cath laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Darki, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meyer G, Vicaut E, Danays T, Agnelli G, Becattini C, Beyer-Westendorf J, Bluhmki E, Bouvaist H, Brenner B, Couturaud F, Dellas C, Empen K, Franca A, Galie N, Geibel A, Goldhaber SZ, Jimenez D, Kozak M, Kupatt C, Kucher N, Lang IM, Lankeit M, Meneveau N, Pacouret G, Palazzini M, Petris A, Pruszczyk P, Rugolotto M, Salvi A, Schellong S, Sebbane M, Sobkowicz B, Stefanovic BS, Thiele H, Torbicki A, Verschuren F, Konstantinides SV; PEITHO Investigators. Fibrinolysis for patients with intermediate-risk pulmonary embolism. N Engl J Med. 2014 Apr 10;370(15):1402-11. doi: 10.1056/NEJMoa1302097. PMID 24716681
- [Background] Kucher N, Boekstegers P, Muller OJ, Kupatt C, Beyer-Westendorf J, Heitzer T, Tebbe U, Horstkotte J, Muller R, Blessing E, Greif M, Lange P, Hoffmann RT, Werth S, Barmeyer A, Hartel D, Grunwald H, Empen K, Baumgartner I. Randomized, controlled trial of ultrasound-assisted catheter-directed thrombolysis for acute intermediate-risk pulmonary embolism. Circulation. 2014 Jan 28;129(4):479-86. doi: 10.1161/CIRCULATIONAHA.113.005544. Epub 2013 Nov 13. PMID 24226805
- [Background] Chatterjee S, Chakraborty A, Weinberg I, Kadakia M, Wilensky RL, Sardar P, Kumbhani DJ, Mukherjee D, Jaff MR, Giri J. Thrombolysis for pulmonary embolism and risk of all-cause mortality, major bleeding, and intracranial hemorrhage: a meta-analysis. JAMA. 2014 Jun 18;311(23):2414-21. doi: 10.1001/jama.2014.5990. PMID 24938564
- [Background] Sharifi M, Bay C, Skrocki L, Rahimi F, Mehdipour M; "MOPETT" Investigators. Moderate pulmonary embolism treated with thrombolysis (from the "MOPETT" Trial). Am J Cardiol. 2013 Jan 15;111(2):273-7. doi: 10.1016/j.amjcard.2012.09.027. Epub 2012 Oct 24. PMID 23102885
- [Background] Zhang Z, Zhai ZG, Liang LR, Liu FF, Yang YH, Wang C. Lower dosage of recombinant tissue-type plasminogen activator (rt-PA) in the treatment of acute pulmonary embolism: a systematic review and meta-analysis. Thromb Res. 2014 Mar;133(3):357-63. doi: 10.1016/j.thromres.2013.12.026. Epub 2013 Dec 23. PMID 24412030
- [Background] Piazza G, Hohlfelder B, Jaff MR, Ouriel K, Engelhardt TC, Sterling KM, Jones NJ, Gurley JC, Bhatheja R, Kennedy RJ, Goswami N, Natarajan K, Rundback J, Sadiq IR, Liu SK, Bhalla N, Raja ML, Weinstock BS, Cynamon J, Elmasri FF, Garcia MJ, Kumar M, Ayerdi J, Soukas P, Kuo W, Liu PY, Goldhaber SZ; SEATTLE II Investigators. A Prospective, Single-Arm, Multicenter Trial of Ultrasound-Facilitated, Catheter-Directed, Low-Dose Fibrinolysis for Acute Massive and Submassive Pulmonary Embolism: The SEATTLE II Study. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1382-1392. doi: 10.1016/j.jcin.2015.04.020. PMID 26315743
- [Background] Tapson VF, Sterling K, Jones N, Elder M, Tripathy U, Brower J, Maholic RL, Ross CB, Natarajan K, Fong P, Greenspon L, Tamaddon H, Piracha AR, Engelhardt T, Katopodis J, Marques V, Sharp ASP, Piazza G, Goldhaber SZ. A Randomized Trial of the Optimum Duration of Acoustic Pulse Thrombolysis Procedure in Acute Intermediate-Risk Pulmonary Embolism: The OPTALYSE PE Trial. JACC Cardiovasc Interv. 2018 Jul 23;11(14):1401-1410. doi: 10.1016/j.jcin.2018.04.008. PMID 30025734
- [Background] Brailovsky, Y. et al. NOVEL BIOMARKERS FOR RISK STRATIFICATION IN ACUTE PULMONARY EMBOLISM. J. Am. Coll. Cardiol. 73, 2088 (2019
- [Background] Part 6: Hemostasis and Thrombosis, Chapter 35: Normal Hemostasis, Fibrinolysis, p. 642-645. Rodak's Hematology. (Saunders, 2020)